## PROTOCOL TITLE:

To examine the effect of Horizant (Gabapentin Enacarbil) in primary Restless Leg Syndrome (RLS) patients who are on Dopaminergic agents and exhibiting Augmentation

## NCT # 02642315

Date of approval: December 8, 2017

## **Statistical Analysis plan:**

Data are analyzed using GraphPad prism software.

Wilcoxon matched-pairs signed rank test used.

Only 1 variable was considered (Augmentation score)

No critical assumptions were made